CLINICAL TRIAL: NCT06302790
Title: Examination of the Acute Effect of Mollii Suit in Children With Cerebral Palsy: A Double-Blind Randomized Controlled Study
Brief Title: Examination of the Acute Effect of Mollii Suit in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Kübra Uğurlu, research assistant, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AcuteMolliiSuitEffects
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Mollii Suit; Cerebral Palsy
Keywords: cerebral palsy; mollii suit; muscle tone; balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The statistician in the study and the physiotherapist performing the evaluation will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Molli Suit Apply Group (Device On) (Active Comparator): Evaluations will be made before the children are dressed in the Mollii Suit, and the evaluations will be repeated after the children are dressed and practiced for 60 minutes.
  Interventions: Other: Molli Suit Apply
- Mollii Suit Placebo Group (Device Off) (Placebo Comparator): Evaluations will be made before the children are dressed in the Mollii Suit, and the evaluations will be repeated after the children are dressed and applied for 60 minutes with the device in off mode.
  Interventions: Other: Molli Suit Apply
- Control Group (No Intervention): Children will be evaluated and the evaluations will be repeated 60 minutes later.

INTERVENTIONS:
Other: Molli Suit Apply — Exopulse Mollii Suit is a neuromodulation application that has been extensively evaluated and is a reliable technique in patients with spasticity. Unlike many neurostimulation techniques that focus only on symptomatic muscles, Suit relieves spasticity and associated pain by stimulating the weakened antagonist of the spastic muscle. Its wearable structure is designed to manage spasticity and associated pain in both upper and lower extremities.
  Arms: Molli Suit Apply Group (Device On); Mollii Suit Placebo Group (Device Off)

SUMMARY:
The aim of our study is to examine the acute effect of Mollii Suit application on balance and muscle tone problems in children with spastic cerebral palsy.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is the most common developmental disorder in childhood. Individuals' independence in daily living activities and participation in education, games, social and community activities are restricted. Technology applications in the field of rehabilitation are gaining momentum. EXOPULSE Mollii Suit method, one of the newest rehabilitation technology products, is a non-invasive neuromodulation approach with a garment that covers the whole body and electrodes placed inside. Designed to improve motor function by reducing spasticity and pain, the method is based on the principle of reciprocal inhibition, which occurs by stimulating the antagonist of a spastic muscle at low frequencies and intensities. Therefore, the aim of our study is to examine the acute effect of Mollii Suit application on balance and muscle tone problems in children with spastic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study
* Having a diagnosis of spastic CP
* 1 or 2 on the Gross Motor Classification System (GMFCS)
* Between the ages of 4-18.

Exclusion Criteria:

* Having GMFCS 3,4,5
* Botulinum Toxin A performed before 3 months or surgical intervention before 6 months
* Having an invasive medical pump (baclofen, insulin, etc.)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | 1 Minute
  Gross Motor Function Classification System (GMFCS) developed by R. Palisano will be used in the classification of motor function.
Modified Tardiue Scale (MTS) | 5 minutes
  The MTS assesses the muscle's response to stretch at given velocities.
Modifiye Modified Ashworth Scale (MAS) | 5 Minutes
  The modified Ashworth scale (MAS), has been applied in clinical practice and research as a measure of spasticity. The modified Ashworth scale purpose is to grade muscle spasticity.
NMC Tests with Seansamove Sensbalance | 5 minutes
  NMC Tests means Neuro Muscular Control tests, and it consists of a number of fully adjustable balance tests. The software calculates up to what point the person is able to perform within the outlines of the exercise, and it will give a score per test. The tests and their duration can be adjusted. Individually applicable and very handy. Once it is adjusted, the same test can be repeated by just pushing a button. Time and results are easy to compare with previous tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rubio-Zarapuz A, Apolo-Arenas MD, Clemente-Suarez VJ, Costa AR, Pardo-Caballero D, Parraca JA. Acute Effects of a Session with The EXOPULSE Mollii Suit in a Fibromyalgia Patient: A Case Report. Int J Environ Res Public Health. 2023 Jan 26;20(3):2209. doi: 10.3390/ijerph20032209. PMID 36767576
- [Result] Pennati GV, Bergling H, Carment L, Borg J, Lindberg PG, Palmcrantz S. Effects of 60 Min Electrostimulation With the EXOPULSE Mollii Suit on Objective Signs of Spasticity. Front Neurol. 2021 Oct 15;12:706610. doi: 10.3389/fneur.2021.706610. eCollection 2021. PMID 34721255
- [Result] Flodstrom C, Viklund Axelsson SA, Nordstrom B. A pilot study of the impact of the electro-suit Mollii(R) on body functions, activity, and participation in children with cerebral palsy. Assist Technol. 2022 Jul 4;34(4):411-417. doi: 10.1080/10400435.2020.1837288. Epub 2021 Mar 29. PMID 33151822
- [Result] Nordstrom B, Prellwitz M. A pilot study of children and parents experiences of the use of a new assistive device, the electro suit Mollii. Assist Technol. 2021 Sep 3;33(5):238-245. doi: 10.1080/10400435.2019.1579267. Epub 2019 Apr 4. PMID 30945989